CLINICAL TRIAL: NCT02731131
Title: A Randomized, Pilot, Open-Label, Monocenter, Efficacy and Safety Study Examining the Effects of Peginterferon Alfa-2a (Pegasys) With or Without Ribavirin (Copegus) in Patients With Chronic Hepatitis D
Brief Title: A Study of Peginterferon Alfa-2a With or Without Ribavirin in Participants With Chronic Hepatitis D (CHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18149
Record Dates: First submitted 2016-04-01; First posted 2016-04-07 (Estimated); Results first posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis D, Chronic
MeSH Terms: conditions — Hepatitis D, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (2):
- Group A: Monotherapy with Peginterferon alfa-2a (Experimental): Participants will receive peginterferon alfa-2a alone, administered over 48 weeks.
  Interventions: Drug: Peginterferon alfa-2a
- Group B: Combination with Peginterferon alfa-2a + Ribavirin (Experimental): Participants will receive combination therapy with peginterferon alfa-2a plus ribavirin, administered over 48 weeks.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a will be administered as 180 micrograms (mcg) once weekly via subcutaneous (SC) injection.
  Other Names: Pegasys
Drug: Ribavirin — Ribavirin will be administered as 1000 to 1200 milligrams (mg) per day in divided oral doses.
  Other Names: Copegus
  Arms: Group B: Combination with Peginterferon alfa-2a + Ribavirin

SUMMARY:
This single-center, randomized, open-label, pilot study is designed to evaluate the efficacy and safety of 48 weeks of treatment with peginterferon alfa-2a alone versus in combination with ribavirin in participants with CHD.

ELIGIBILITY:
Inclusion Criteria:

* Positive hepatitis B surface antigen (HBsAg) for the prior 6 months
* Positive anti-delta for the prior 3 months
* Positive HDV RNA at Screening
* Elevated ALT (1 to 10 times upper limit of normal) prior to first dose
* Chronic, necroinflammatory hepatitis documented within the prior 18 months (non-cirrhotic) or 30 months (cirrhotic)
* Negative pregnancy and adequate contraceptive use

Exclusion Criteria:

* Antiviral therapy for CHD within previous 3 months
* Positive for hepatitis A or C, or human immunodeficiency virus (HIV)
* Increased risk of metabolic liver disease
* Decompensated liver disease
* Elevated bilirubin
* Poor hematologic or renal function
* Drug/alcohol abuse within 1 year prior to study
* History of significant psychiatric, autoimmune, pulmonary, cardiac, oncologic, or thyroid disease
* Organ transplantation with existing functional graft
* Retinopathy or other ophthalmologic complication of diabetes or hypertension
* Inclusion in another investigational trial within previous 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (1):
- Cagliari, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Monotherapy With Peginterferon Alfa-2a: Participants received peginterferon alfa-2a for 48 weeks as 180 micrograms (mcg) once weekly via subcutaneous (SC) injection.
- Group B: Combination With Peginterferon Alfa-2a + Ribavirin: Participants received peginterferon alfa-2a plus ribavirin for 48 weeks. Peginterferon alfa-2a was given as 180 mcg once weekly via SC injection. Ribavirin was administered as 1000 to 1200 milligrams (mg) per day in divided (morning/evening) oral doses. The specific dose was determined according to the participant's body weight at Baseline.
Period: Overall Study
Arm/Group | Group A: Monotherapy With Peginterferon Alfa-2a | Group B: Combination With Peginterferon Alfa-2a + Ribavirin
Started | 6 | 6
Completed | 6 | 4
Not Completed | 0 | 2
Not completed — Psychiatric Disorder | 0 | 1
Not completed — Refused Therapy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All participants who received at least one dose of study medication.
Groups:
- Group A: Monotherapy With Peginterferon Alfa-2a: Participants received peginterferon alfa-2a for 48 weeks as 180 mcg once weekly via SC injection.
- Group B: Combination With Peginterferon Alfa-2a + Ribavirin: Participants received peginterferon alfa-2a plus ribavirin for 48 weeks. Peginterferon alfa-2a was given as 180 mcg once weekly via SC injection. Ribavirin was administered as 1000 to 1200 mg per day in divided (morning/evening) oral doses. The specific dose was determined according to the participant's body weight at Baseline.
- Total: Total of all reporting groups
Arm/Group | Group A: Monotherapy With Peginterferon Alfa-2a | Group B: Combination With Peginterferon Alfa-2a + Ribavirin | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (9.2) | 49.2 (7.4) | 48.2 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Alanine Aminotransferase (ALT) Normalization Plus Negative Hepatitis D Virus (HDV) Ribonucleic Acid (RNA) at 48 Weeks After End of Treatment
Description: Normalized ALT was defined as ALT value above the upper limit of normal (ULN) at Baseline with a decrease in ALT value to at/below the ULN at 48 weeks after end of treatment (Week 96). Negative HDV RNA was defined as HDV RNA not detected by polymerase chain reaction (PCR). The number of participants with ALT normalization and negative HDV RNA at Week 96 was reported.
Time Frame: Week 96
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Group A: Monotherapy With Peginterferon Alfa-2a | Group B: Combination With Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 6 | 6
participants | 0 | 1
Statistical Analysis 1: Comparison: Group A: Monotherapy With Peginterferon Alfa-2a vs Group B: Combination With Peginterferon Alfa-2a + Ribavirin; Test type: Superiority or Other; p = 0.30, Fisher Exact

2. Secondary Outcome: Number of Participants With ALT Normalization Plus Negative HDV RNA at End of Treatment
Description: Normalized ALT was defined as ALT value above the ULN at Baseline with a decrease in ALT value to at/below the ULN at the end of treatment (Week 48). Negative HDV RNA was defined as HDV RNA not detected by PCR. The number of participants with ALT normalization and negative HDV RNA at Week 48 was reported.
Time Frame: Week 48
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Group A: Monotherapy With Peginterferon Alfa-2a | Group B: Combination With Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 6 | 6
participants | 0 | 0

3. Secondary Outcome: Number of Participants With ALT Normalization at 48 Weeks After End of Treatment
Description: Normalized ALT was defined as ALT value above the ULN at Baseline with a decrease in ALT value to at/below the ULN at 48 weeks after end of treatment (Week 96). The number of participants with ALT normalization at Week 96 was reported.
Time Frame: Week 96
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Group A: Monotherapy With Peginterferon Alfa-2a | Group B: Combination With Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 6 | 6
participants | 3 | 1
Statistical Analysis 1: Comparison: Group A: Monotherapy With Peginterferon Alfa-2a vs Group B: Combination With Peginterferon Alfa-2a + Ribavirin; Test type: Superiority or Other; p = 0.22, Fisher Exact

4. Secondary Outcome: Number of Participants With ALT Normalization at End of Treatment
Description: Normalized ALT was defined as ALT value above the ULN at Baseline with a decrease in ALT value to at/below the ULN at the end of treatment (Week 48). The number of participants with ALT normalization at Week 48 was reported.
Time Frame: Week 48
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Group A: Monotherapy With Peginterferon Alfa-2a | Group B: Combination With Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 6 | 6
participants | 1 | 0
Statistical Analysis 1: Comparison: Group A: Monotherapy With Peginterferon Alfa-2a vs Group B: Combination With Peginterferon Alfa-2a + Ribavirin; Test type: Superiority or Other; p = 0.30, Fisher Exact

5. Secondary Outcome: Number of Participants With Negative HDV RNA at 48 Weeks After End of Treatment
Description: Negative HDV RNA was defined as HDV RNA not detected by PCR. The number of participants with negative HDV RNA at 48 weeks after end of treatment (Week 96) was reported.
Time Frame: Week 96
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Group A: Monotherapy With Peginterferon Alfa-2a | Group B: Combination With Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 6 | 6
participants | 0 | 1
Statistical Analysis 1: Comparison: Group A: Monotherapy With Peginterferon Alfa-2a vs Group B: Combination With Peginterferon Alfa-2a + Ribavirin; Test type: Superiority or Other; p = 0.30, Fisher Exact

6. Secondary Outcome: Number of Participants With Negative HDV RNA at End of Treatment
Description: Negative HDV RNA was defined as HDV RNA not detected by PCR. The number of participants with negative HDV RNA at the end of treatment (Week 48) was reported.
Time Frame: Week 48
Population: ITT Population.
Measure: Number; unit: participants
Arm/Group | Group A: Monotherapy With Peginterferon Alfa-2a | Group B: Combination With Peginterferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 6 | 6
participants | 1 | 2
Statistical Analysis 1: Comparison: Group A: Monotherapy With Peginterferon Alfa-2a vs Group B: Combination With Peginterferon Alfa-2a + Ribavirin; Test type: Superiority or Other; p = 0.50, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline through 24 weeks after end of treatment (up to 72 weeks)
Description: Safety Population: All randomized participants who received at least one dose of study medication and had at least one post-baseline safety assessment.
Arm/Group | Group A: Monotherapy With Peginterferon Alfa-2a | Group B: Combination With Peginterferon Alfa-2a + Ribavirin
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Monotherapy With Peginterferon Alfa-2a (N=6) | Group B: Combination With Peginterferon Alfa-2a + Ribavirin (N=6)
Asthenia (General disorders) | 5 | 3
Pyrexia (General disorders) | 5 | 3
Influenza like illness (General disorders) | 2 | 1
Malaise (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 3
Depression (Psychiatric disorders) | 2 | 3
Irritability (Psychiatric disorders) | 2 | 3
Emotional disorder (Psychiatric disorders) | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Conjunctivitis (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.